CLINICAL TRIAL: NCT02142933
Title: 1) Accuracy of the Vagino-perineal Versus the Standard Dual Swab for Detection of Group B Streptococcus in Pregnancy 2) Prevalence and Risk Factors of Extended-Spectrum Beta-Lactamase Producing Enterobacteriaceae in Pregnancy
Brief Title: Simplified GBS Screening and Prevalence of ESBL in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Stiftung Forschung Infektionskrankheiten, Basel, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EKNZ-2014-087
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Group B Streptococcal Infection; Infection Due to ESBL Bacteria
Keywords: colonization; screening; group B streptococci; extended-spectrum beta-lactamase; enterobacteriaceae
MeSH Terms: conditions — Streptococcal Infections

ARMS (1):
- rectal swab and vagino-perineal swab (Other): single-arm
  Interventions: Other: vagino-perineal swab

INTERVENTIONS:
Other: vagino-perineal swab

SUMMARY:
1. At the University Hospital Basel, Switzerland, a simplified screening for group B streptococci (GBS) of vagina and perineum has been performed since several years. Reliable detection of GBS is critical to prevent GBS transmission during delivery with antimicrobial prophylaxis. Transmission of GBS to the neonate may otherwise lead to severe infection and complications in the neonate. Centers for Disease Control and Prevention (CDC) and other international organizations recommend a vaginal and additional rectal swab.We therefore aim to test this simplified screening against the international gold standard.
2. Antibiotic resistant bacteria may reside in the genital tract of an expected mother and may be transmitted to the new-born during delivery. In case of infection of the pregnant woman or the neonate, application of standard antimicrobial treatment will insufficiently cover these extended spectrum beta-lactamase (ESBL) producing bacteria. Therefore, colonization with ESBL in pregnancy needs to be known to potentially deliver adequate antimicrobial treatment.

DETAILED DESCRIPTION:
Transmission of GBS under delivery leads in 1/1000 of live births to severe sepsis in the neonate and may have serious sequelae including death. Most of the cases concern early onset sepsis which occurs in the first three to seven days after birth. Several randomized studies showed that antibiotic prophylaxis during delivery reduces the risk of early onset sepsis in the neonate in 85%, whereas late onset sepsis was not affected. Accurate screening including appropriate culture methods are critical for the wealth of the newborn and the decision regarding application of antibiotic prophylaxis to the mother. In this study we compare a simplified test algorithm taking swabs from the vagina and the perineum only versus a combined vaginal and rectal swab for GBS culture which is the current gold standard of diagnosis as the culture yield for GBS increases substantially when samples are taken from both the lower vagina and the rectum compared to swabbing the vagina or endocervix only. There is certain reluctance for performing a rectal swab as it has been associated with discomfort.

The study aims to demonstrate that this simplified vagino-perineal swab leads to a similar GBS detection rate as compared to the gold standard comprising of a combined vaginal and rectal swab. We further aim to systematically assess the degree of discomfort with the rectal swab and compare the costs when applying those different methods.

Additionally we aim to determine the prevalence and risk factors of community acquired ESBL by further processing the swabs in the appropriate culture media and filling in a standardized questionnaire.

We plan a prospective cohort study with inclusion of 450 pregnant women who attend the outpatient obstetric clinic for routine control in the third trimester.

ELIGIBILITY:
Inclusion Criteria:

* third trimester pregnancy
* must attend clinic for routine screening for group B streptococcus (GBS)

Exclusion Criteria:

* detection of group B streptococcus in urine
* history of neonatal group B streptococcal sepsis in previous pregnancy
* antibiotic treatment within the past 2 weeks before routine GBS screening
* delivery < 37 gestational week
* condition or disorders suggestive for urinary tract infection, genital tract infection, or bacterial vaginosis
* language barrier (insufficient knowledge of German or English)
* the expected mother has any other condition, that, in the opinion of the investigator or treating physician, would jeopardize the safety or rights of the expected mother participating in the study, or would confound the results of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Presence of group B streptococci in genital tract | third trimester of pregnancy
  on routine visit in third trimester of pregnancy
Presence of colonizing extended-spectrum beta-lactamase enterobacteriaceae in genital tract | third trimester of pregnancy
  on routine visit in third trimester pregnancy

SECONDARY OUTCOMES:
Evaluation of pain during performance of rectal swab | third trimester of pregnancy
  On routine visit in third trimester pregnancy
Evaluation of discomfort during performance of rectal swab | third trimester of pregnancy
  On routine visit in third trimester pregnancy
Evaluation of stress during performance of rectal swab | third trimester of pregnancy
  On routine visit in third trimester pregnancy
risk factors for ESBL carriage | third trimester of pregnancy
  on routine visit in third trimester of pregnancy

OTHER OUTCOMES:
Evaluation of costs for additional rectal swab | between 38 and 42 gestational week
  On routine visit in third trimester pregnancy
Resistance pattern of ESBL bacteria | between 38 and 42 gestational week

CONTACTS AND LOCATIONS:
Overall Officials: Irene Hoesli, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland